CLINICAL TRIAL: NCT02035826
Title: A Randomized Trial of Patient Financial Incentives to Reduce CVD Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Harvard Vanguard Medical Associates (Other); Geisinger Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2013P001902/BWH
Record Dates: First submitted 2014-01-10; First posted 2014-01-14 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2013-11

CONDITIONS: Cardiovascular Disease (CVD)
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1 (Active Comparator): Arm (Expected Value) 2 Digit Match 1st Digit Match 2nd Digit Match Arm 1 ($2.80) $100 $10 $10
  Interventions: Behavioral: Behavioral Economics Intervention
- Arm 2 (Active Comparator): Arm (Expected Value) 2 Digit Match 1st Digit Match 2nd Digit Match Arm 2 ($1.40) $50 $5 $5
  Interventions: Behavioral: Behavioral Economics Intervention
- Arm 3 (Active Comparator): Arm (Expected Value) 2 Digit Match 1st Digit Match 2nd Digit Match Arm 3 ($0.70) $25 $5 $0
  Interventions: Behavioral: Behavioral Economics Intervention
- Arm 4 (No Intervention): Control Arm

INTERVENTIONS:
Behavioral: Behavioral Economics Intervention — Patients will receive an active intervention for 3 months followed by 3 months of observation. Incentives will be awarded at the end of the first 3 months, based on an improvement of at least 10 mg/dl in LDL relative to the patient's baseline LDL or achieving or sustaining LDL of 100, depending on baseline LDL and FRS. Adherence in all groups will be measured using Vitality GlowCaps as a recording device. Patients in all arms will be given the GlowCaps and instructions on use. Patients will receive adherence feedback electronically with daily lottery awards to match the timing of their task.
  Arms: Arm 1; Arm 2; Arm 3

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of death in the United States. Despite strong evidence that reducing low-density lipoproteins (LDL) with statins successfully lowers CVD risk, physicians under-prescribe statins, physicians fail to intensify treatment when indicated, and more than 50% of patients stop taking statins within one year of ﬁrst prescription though such therapy typically should be life-long. In this study, we will test the effectiveness of different financial incentives in increasing statin use and reducing LDL cholesterol among patients with poor cholesterol control who are at very high risk for CVD. The application of conceptual approaches from behavioral economics offers considerable promise in advancing health and health care. We will test these approaches among patients at very high risk of CVD at Harvard Vanguard Medical Associates. Using a 4-arm, cluster-randomized controlled trial, we aim to answer these questions: [1] How does the provision of patient incentives compare to no incentives at all? [2] Is success with patient incentives improved by increasing the financial amounts? [3] Are results sustained after incentives and other interventions are withdrawn?

Study Objectives and Hypothesis

Aim 1: To evaluate the effectiveness of varying patient incentives on improvement in LDL cholesterol relative to usual care during a 3-month intervention among patients at high risk of CVD. H1: Each of the incentives will be more effective than usual care in reducing LDL cholesterol.

Aim 2: To evaluate the relative effectiveness of those intervention arms superior to control in reducing LDL cholesterol. H2: Higher incentive amounts for patients will be more effective than lower incentive amounts.

Aim 3: To evaluate the impact of each effective intervention in sustaining adherence and reduced LDL after the 3-month intervention period.

Aim 4: To conduct a rigorous process evaluation to examine why some incentives were more effective than others and to address other factors relevant to broader implementation.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-80 yrs
* FRS of > 20% with LDL > 120, or FRS = 10-20% with LDL > 140, or a coronary artery disease equivalent (diabetes, peripheral artery disease, ischemic CVD, arteriosclerotic CVD, stroke/TIA, CABG, coronary stenting, or coronary bypass anastomosis) with LDL > 120.

Exclusion Criteria:

* Patients with a history of side effects to statins. Patients with a history of side effects to statins will be forwarded to the study's medical monitor (a physician aligned with the study) and may still participate in the study if, after the medical monitor reviews the patient's medical record, he/she determines that the patient may safely participate in the study;
* Patients who will not or cannot give consent;
* Patients with terminal illness who are no longer suitable candidates for aggressive lipid management as determined by the patient's primary care physician;
* Patients with ALT values detected at greater than 80 U/L;
* Patients with active or progressive liver disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
LDL Cholesterol | Baseline and 3 months
  The primary outcome will be change in LDL between baseline (prior to randomization) and 3 months.

SECONDARY OUTCOMES:
LDL Cholesterol | Baseline to 6 months
  We will measure change in LDL from baseline to 6 months.

OTHER OUTCOMES:
Hemoglobin A1c | Baseline and 3 months
  We will also measure Hemoglobin A1c, an assessment of intermediate term glycemic control, among patients with diabetes. This measure is related to CVD risk but is not a target of the intervention. We measure it to examine positive or negative spillover effects from targeting LDL cholesterol: a focus on LDL may crowd out attention to other conditions or, alternatively, might stimulate it.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Issac, MD, MPH, Principal Investigator — Harvard Vanguard Medical Associates
Locations (1):
- Harvard Vanguard Medical Associates, Boston, Massachusetts, United States